CLINICAL TRIAL: NCT02621684
Title: A Pilot Study of Physical Activity Intervention in African American Men After Radical Prostatectomy
Brief Title: Physical Activity Intervention in African American Men After Radical Prostatectomy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not able to enroll any participants due to disinterest
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 201410072
Record Dates: First submitted 2015-11-25; First posted 2015-12-03 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2016-01

CONDITIONS: Prostatectomy; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1: Aerobics (Experimental): * Complete baseline questionnaires either online or on paper
  * Questionnaires will also be completed at 6 weeks, 12 weeks, and 16 weeks after baseline
  * Participants will be asked to wear an accelerometer for 7 days at baseline, 12 weeks, and 16 weeks.
  * Receive printed materials from the American Cancer Society about cancer management and standard physical activity recommendations.
  * Require physical evaluation and orientation to the WellAware gym
  * 12 week walking program at the WellAware Center
    * required to check in with gym staff to check attendance
    * advised to walk at own pace for 3 days per week
    * 15 minutes per day for the first 2 weeks
    * 30 minutes per day for the next 2 weeks
    * 50 minutes or more for remaining weeks
  Interventions: Other: Community Health Activities Model Program for Seniors (CHAMPS); Other: Lifetime Total Physical Activity Questionnaire; Other: Expanded Prostate Cancer Index Composite (EPIC); Other: International Physical Activity Prevalence Study Environmental Module; Other: Godin Leisure-Time Exercise Questionnaire (GLTEQ); Other: Questionnaire regarding behavior/lifestyle changes since diagnosis; Other: 12 week Walking Program
- Arm 2: Resistance training (Experimental): * Complete baseline questionnaires either online or on paper
  * Questionnaires will also be completed at 6 weeks, 12 weeks, and 16 weeks after baseline
  * Participants will be asked to wear an accelerometer for 7 days at baseline, 12 weeks, and 16 weeks.
  * Receive printed materials from the American Cancer Society about cancer management and standard physical activity recommendations.
  * Require physical evaluation and orientation to the WellAware gym
  * 12 week weight lifting program at WellAware Center
    * exercise physiologists will work with each patient to develop a custom routine
    * exercise load will start at 60% of one-repetition maximum and progress from 8 to 12 repetitions
    * 2-4 sets of repetition exercises will be performed to target upper & lower muscle groups
    * resistance load will be added by 5 pounds when patients can complete more than 12 repetitions
  Interventions: Other: Community Health Activities Model Program for Seniors (CHAMPS); Other: Lifetime Total Physical Activity Questionnaire; Other: Expanded Prostate Cancer Index Composite (EPIC); Other: International Physical Activity Prevalence Study Environmental Module; Other: Godin Leisure-Time Exercise Questionnaire (GLTEQ); Other: Questionnaire regarding behavior/lifestyle changes since diagnosis; Other: 12 week Resistance Training Program
- Arm 3: Usual care (Active Comparator): * Complete baseline questionnaires either online or on paper
  * Questionnaires will also be completed at 6 weeks, 12 weeks, and 16 weeks after baseline
  * Participants will be asked to wear an accelerometer for 7 days at baseline, 12 weeks, and 16 weeks.
  * Receive printed materials from the American Cancer Society about cancer management and standard physical activity recommendations.
  Interventions: Other: Community Health Activities Model Program for Seniors (CHAMPS); Other: Lifetime Total Physical Activity Questionnaire; Other: Expanded Prostate Cancer Index Composite (EPIC); Other: International Physical Activity Prevalence Study Environmental Module; Other: Godin Leisure-Time Exercise Questionnaire (GLTEQ); Other: Questionnaire regarding behavior/lifestyle changes since diagnosis

INTERVENTIONS:
Other: Community Health Activities Model Program for Seniors (CHAMPS) — * Physical activity questionnaire for older adults
  * Asks about activities in the past 4 weeks
  * 41 questions and asks to notate how long the activity took
Other: Lifetime Total Physical Activity Questionnaire — * Questions about leisure time (27) and household activities (5)
  * Mark if participated in the activity during the past year, ages 51-65, 35-50, 23-34, and onset of puberty through 21 years
Other: Expanded Prostate Cancer Index Composite (EPIC) — * Measures urinary and sexual function before and after prostate cancer treatment
  * 7 questions about urinary function
  * 9 questions about sexual function
Other: International Physical Activity Prevalence Study Environmental Module — -The 17-item Physical Activity Neighborhood Environment Scale can be used to assess the environmental factors for walking and bicycling in various neighborhoods.
Other: Godin Leisure-Time Exercise Questionnaire (GLTEQ) — -4 item query of usual leisure time exercise habits
Other: Questionnaire regarding behavior/lifestyle changes since diagnosis
Other: 12 week Walking Program
  Arms: Arm 1: Aerobics
Other: 12 week Resistance Training Program
  Arms: Arm 2: Resistance training

SUMMARY:
The purpose of this pilot study is to evaluate the feasibility of recruiting African American prostate cancer survivors to a 12 week physical activity intervention study of three arms (aerobics, resistance training, and usual care) through physician referral and community advertisement strategies. In addition, the investigators will investigate the acceptance rate of the intervention and gather preliminary results on the effect of exercise on African American men's urinary and sexual functions. These data can then be used to refine the intervention and its implementation model, and to inform the submission of a larger grant to the National Institutes of Health.

ELIGIBILITY:
Inclusion Criteria:

* Speaks English
* African American
* Radical prostatectomy for treatment of prostate cancer within the past 12 months
* Cleared by physician to safely participate in a physical exercise program

Exclusion Criteria:

* Does not speak English
* Non-African American
* Previously undergone radiation treatment to the pelvis
* Previously undergone major pelvic surgery
* Known urethral stricture, colostomy, or inability to urinate requiring chronic urinary catheter

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-11; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate comparisons between physician referral and community advertisement | Completion of study (approximately 3.5 years)
Attrition rate in each arm | Completion of study (approximately 3.5 years)
  * Evaluate percentage of finished duration of walking in each session and percentage of total finished session in the aerobic exercise arm.
  * Evaluate the percentage of attended sessions in the resistance training arm
Intervention effectiveness as measured by change in accelerometer measured physical activity | Completion of study (approximately 3.5 years)
Intervention effectiveness as measured by change in self-reported urinary/sexual function as measured by Expanded Prostate Cancer Index Composite (EPIC) | Completion of study (approximately 3.5 years)
  -Intervention effectiveness will be compared between the three arms by comparing the change in self-reported urinary and sexual function. Mixed effects regression will be used to account for the longitudinal design.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Yang, Ph.D., Principal Investigator — Washington University School of Medicine

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu